CLINICAL TRIAL: NCT01449266
Title: Safety and Dialysability of Dotarem® in Dialysed Patients - Phase 1 Clinical Study
Brief Title: Safety and Dialysability of Dotarem® in Dialysed Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DGD-44-054
Record Dates: First submitted 2011-10-03; First posted 2011-10-10 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: End-stage Renal Failure
Keywords: Dotarem; Dialyses; Dialysed; Safety; Safety and dialysability of Dotarem in dialysed patients
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dotarem®-injected patients (Other): Male or female subjects, aged ≥18 years,suffering from end-stage renal failure and requiring hemodialysis treatment 3 times per week, were submitted to a single Dotarem® IV injection at 0.1 mmol/kg before being submitted to 3 hemodialysis sessions to assess the decrease of Dotarem® concentration in the blood.
  Interventions: Drug: Dotarem® IV injection at 0.1 mmol/kg

INTERVENTIONS:
Drug: Dotarem® IV injection at 0.1 mmol/kg — Dotarem® was IV administered at a dose of 0.1 mmoL/kg (0.2 mL/kg).
  Other Names: gadoterate meglumine; gadoteric acid

SUMMARY:
To evaluate the dialysability of Dotarem®, after an IV injection of 0.1 mmol/kg in patients with chronic renal failure who require hemodialysis treatment.

DETAILED DESCRIPTION:
Ten adult patients suffering from end stage renal failure and requiring hemodialysis treatment for 3 times were enrolled. Patients received a single dose of Dotarem® at 0.1 mmol/kg before being submitted to hemodialysis to assess the dialysability of Dotarem® . After injection of Dotarem®, 3 sessions of hemodialysis were performed as follows:

The first hemodialysis session started between 1 to 2 h after the injection; The second hemodialysis session occurred 2 days (i.e., 48 ± 2 h) after the Dotarem® injection; The third hemodialysis session occurred 4 days (i.e., 96 ± 4 h) after the Dotarem® injection.

The decrease in serum Dotarem® concentration was assessed after each hemodialysis session. Safety assessments included adverse events (AEs), vital signs, injection-site tolerance, and laboratory assessments.Two safety follow-up visits were performed: one 3 weeks (± 2 days) and one 3 months (± 4 days) after the Dotarem® injection.

ELIGIBILITY:
Inclusion Criteria:

Male or female, aged ≥18 years

* Subjects suffering from end-stage renal failure who require hemodialysis treatment for 3 times per week (or equivalent to allow overnight dialysis being rescheduled as appropriate per protocol)
* Female Subjects with effective contraception (contraceptive pill or Intra-Uterine Device), or surgically sterilized or post-menopausal (minimum 12 months amenorrhea)
* Subjects having provided their written informed consent to participate in the trial

Exclusion Criteria:

* Known allergy to gadolinium chelates
* Pregnant, breast feeding, or planning to become pregnant during the trial
* Having received or scheduled to be injected with any contrast agent within 7 days before or after the Dotarem® injection
* Schedule to receive erythropoietin (EPO) or iron therapy during 1 week after the Dotarem® injection
* Evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Evidence of hepatitis C and/or positive hepatitis C antibody and/or positive hepatitis B surface antigen
* History of hypersensitivity to drugs with a similar chemical structure

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Mesens, MD, Principal Investigator — Clinical Pharmacology Unit Antwerp, Belgium
Locations (1):
- Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Dotarem® Injected Patients: Male or female, aged ≥18 years
  • Subjects suffering from end-stage renal failure who require hemodialysis treatment for 3 times per week (or equivalent to allow overnight dialysis being rescheduled as appropriate per protocol)
  Dotarem®: Dotarem® was administered at a dose of 0.1 mmoL/kg (0.2 mL/kg).
Period: Overall Study
Arm/Group | Dotarem® Injected Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No statistical calculation of sample size was done. According to the literature, a sample of 10 patients was judged sufficient to evaluate the dialysability of Dotarem®.
Groups:
- Dotarem®-Injected Patients: Male or female, aged ≥18 years
  • Subjects suffering from end-stage renal failure who require hemodialysis treatment for 3 times per week (or equivalent to allow overnight dialysis being rescheduled as appropriate per protocol)
  Dotarem®: Dotarem® was administered at a dose of 0.1 mmoL/kg (0.2 mL/kg).
Arm/Group | Dotarem®-Injected Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 64.0 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  Belgium | 10

OUTCOME MEASURES:

1. Primary Outcome: Dialysability of Dotarem® in Dialysed Patients
Description: To evaluate the decrease in seric concentration of gadolinium, after each hemodialysis session of patients injected with 0.1 mmol/kg of Dotarem® . The percent change of gadolinium concentration is calculated by estimating the amount of serum gadolinium before and after each hemodialysis session. Calculations are performed only for subjects with concentration above the lower limit of quantification (LLQ)
Time Frame: Dotarem® dialysability assessed up to 4 days after Dotarem® administration
Population: After second hemodialysis, 3 subjects had Gd concentration<LLQ and are not included in the analysis; after third hemodialysis, 8 subjects had Gd concentration<LLQ and are not included in the analysis
Measure: Geometric Mean (Full Range); unit: percent change in Gd concentration
Groups:
- Dotarem® Injected Patients: Male or female, aged ≥18 years
  • Subjects suffering from end-stage renal failure who require hemodialysis treatment for 3 times per week (or equivalent to allow overnight dialysis being rescheduled as appropriate per protocol)
Arm/Group | Dotarem® Injected Patients
Number analyzed (Participants) | 10
percent change in Gd concentration
  Percent change at 0.5h after first hemodialysis | -88.2 [-93.5 to -84.7]
  Percent change at 1.5h after first hemodialysis | -93.4 [-95.7 to -90.3]
  Percent change at 4h after first hemodialysis | -97.1 [-99.1 to -90.5]
  Percent change at 4h after second hemodialysis n=7 | -94.8 [-97.7 to -84.8]
  Percent change at 4h after third hemodialysis n=2 | -89.9 [-94.9 to -85.0]

2. Secondary Outcome: Safety of Dotarem® in Dialysed Patients Evaluated by the Number of Patients Experiencing Adverse Events.
Description: To evaluate the biological and clinical safety of Dotarem® by assessing vital signs, biological parameters, injection-site tolerance, through a 4-day post injection follow-up, adverse events through a 3-week post injection period and serious adverse events through a 3-month post injection period.
Time Frame: Safety assessed from patients inclusion until the last follow-up visit 3 months after Dotarem® administration
Measure: Number; unit: participants
Arm/Group | Dotarem® Injected Patients
Number analyzed (Participants) | 10
participants | 8

3. Post Hoc Outcome: Percent Change in Gadolinium Serum Concentration 4h After Second Hemodialysis Session, Estimated From Subjects With Concentration Data Above the Limit of Detection
Description: Evaluation of the decrease in seric concentration of gadolinium, 4h after the second hemodialysis session of patients injected with 0.1 mmol/kg of Dotarem®. The percent change of gadolinium concentration was estimated from the concentration of gadolinium after Dotarem® injection. Only subjects with gadolinium concentration above the lower limit of quantification (LLQ) were kept for analysis.
Time Frame: Dotarem® dialysability assessed 4h after second hemodialysis session which took place 2 days after Dotarem® administration
Population: 3 subjects had a gadolinium concentration <LLQ after the second hemodialysis session
Measure: Geometric Mean (Full Range); unit: Percent change in Gd concentration
Arm/Group | Dotarem® Injected Patients
Number analyzed (Participants) | 7
Percent change in Gd concentration | -99.5 [-99.8 to -98.6]

4. Post Hoc Outcome: Percent Change in Gadolinium Serum Concentration 4h After Third Hemodialysis Session, Estimated From Subjects With Concentration Data Above the Limit of Detection
Description: The evaluation of the decrease in seric concentration of gadolinium, 4h after the third hemodialysis session of patients injected with 0.1 mmol/kg of Dotarem®. The percent change of gadolinium concentration was estimated from the concentration of gadolinium after Dotarem® injection. Only subjects with gadolinium concentration above the lower limit of detection were kept for analysis.
Time Frame: Dotarem® dialysability assessed 4h after third hemodialysis session which took place 4 days after Dotarem® administration
Population: 8 subjects had a gadolinium concentration <LLQ after third hemodialysis session
Measure: Geometric Mean (Full Range); unit: percent change in Gd concentration
Arm/Group | Dotarem® Injected Patients
Number analyzed (Participants) | 2
percent change in Gd concentration | -99.7 [-99.8 to -99.7]

ADVERSE EVENTS:
Time Frame: Safety assessment was performed at the day 1, day 2, and day 4 after Dotarem® injection. Two safety follow-up visits were performed at 3 weeks (+/- 2 days) and at 3 months (+/- 4 days) after Dotarem® injection.
Description: Adverse events (AEs) were followed from the subject's screening to the first safety follow-up visit (3 weeks +/- 2 days after the Dotarem® injection). At the second safety follow-up visit (3 months +/- 4 days after the Dotarem® injection), only Serious Adverse Events (SAEs) were evaluated.
Groups:
- Dotarem® Injected Patients: Male or female, aged ≥18 years
  • Subjects suffering from end-stage renal failure who require hemodialysis treatment for 3 times per week (or equivalent to allow overnight dialysis being rescheduled as appropriate per protocol)
  Dotarem: Dotarem® was administered at a single dose of 0.1 mmoL/kg (0.2 mL/kg).
Arm/Group | Dotarem® Injected Patients
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem® Injected Patients (N=10)
moderate sepsis (Infections and infestations) | 2 (2) — Five days after Dotarem® injection subject experienced moderate sepsis deemed not related. Subject was hospitalized and recovered after 15 days following antibiotic treatment. This AE was considered as not related to the Dotarem® injection.
severe respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
severe peripheral ischemia (Vascular disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
moderate thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
severe urosepsis (Infections and infestations) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Dialysis device insertion (Surgical and medical procedures) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Nephrectomy (Surgical and medical procedures) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem® Injected Patients (N=10)
Hypotension (Vascular disorders) | 5 (5) — This adverse event was considered as not related to the Dotarem® injection.
Headache (Nervous system disorders) | 3 (3) — This adverse event was considered as not related to the Dotarem® injection.
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) — This adverse event was considered as not related to the Dotarem® injection.
Anemia (Blood and lymphatic system disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Abdominal pain (Gastrointestinal disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
influenza-like illness (General disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
thirst (General disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Dizziness postural (Nervous system disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Presyncope (Nervous system disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.
Hypertension (Vascular disorders) | 1 (1) — This adverse event was considered as not related to the Dotarem® injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished data given to the investigator may be transmitted to a third party without approval by the sponsor. The data are the exclusive property of Guerbet.

The investigator undertakes to submit to Guerbet any articles or papers related to this study within 30 days of their submission to journals or congresses.

All publications must have the joint agreement of the investigator and the sponsor.

The investigator remains independent with no relationship of subordination with Guerbet.